CLINICAL TRIAL: NCT04213287
Title: Evaluation of Multimodal Analgesia Methods in Patients Who Underwent IPACK Block in Total Knee Arthroplasty
Brief Title: Multimodal Analgesia Methods in Patients Undergoing IPACK Block in Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara Diskapi Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ilkay baran akkuş, Principal Investigator, Ankara Diskapi Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 70/13
Record Dates: First submitted 2019-12-23; First posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: IPACK Block Multimodal Analgesia; Postoperative NRS Scores
MeSH Terms: interventions — dexketoprofen trometamol; Anesthesia, Spinal

STUDY DESIGN:
Intervention Model Description: Power analysis will be done after a pilot study. Number of patient may vary.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peri-Articular Injections and IPACK (Experimental): Spinal anesthetic with 2,5 ml 0,5% heavy bupivacaine
  At the end of surgery;
  PAI: 30 ml 0,025% bupivacaine and
  IPACK: 20 ml 0,025% bupivacaine
  Interventions: Drug: Dexketoprofen Trometamol; Other: spinal anesthesia; Other: IPACK; Other: PAI
- Adductor Canal Block, and IPACK (Active Comparator): Spinal anesthetic with 2,5 ml 0,5% heavy bupivacaine
  At the end of surgery;
  ADD: 20 ml 0,025% bupivacaine and
  IPACK: 20 ml 0,025% bupivacaine
  Interventions: Drug: Dexketoprofen Trometamol; Other: spinal anesthesia; Other: IPACK; Other: Adductor canal block

INTERVENTIONS:
Drug: Dexketoprofen Trometamol — Drug: Dexketoprofen Trometamol oral tablet
Other: spinal anesthesia — Drug: heavy bupivacaine 2,5 ml 0,5%
Other: IPACK — Drug: bupivacaine 20 ml 0,025%
Other: PAI — Drug: bupivacaine 30 ml 0,025%
  Arms: Peri-Articular Injections and IPACK
Other: Adductor canal block — Drug: bupivacaine 20 ml 0,025%
  Arms: Adductor Canal Block, and IPACK

SUMMARY:
A comparison of two pain control methods - the combination of Adductor Canal Block (ACB)/Infiltration of the interspace between the popliteal artery and the capsule of the posterior knee (IPACK) versus the Periarticular Injection (PAI)/ Infiltration of the interspace between the popliteal artery and the capsule of the posterior knee (IPACK) - in patients undergoing total knee arthroplasty. dexketoprofen and paracetamol will be added to both groups and multimodal analgesia will be applied. Primary outcome is NRS pain scores with ambulation on postoperative day one (24 hours post-block administration).

DETAILED DESCRIPTION:
Postoperative pain after total knee arthroplasty is serious and difficult to management. Multimodal analgesia recommended for the pain management. For these reasons, we planned a study involving two multimodal analgesia regimens. Patients who will undergo total knee arthroplasty will receive preemptive oral analgesic (dexketofrofen) 1 hour before the operation. Surgery will be initiated after spinal anesthesia is applied to the patients. Two pain control methods - the combination of Adductor Canal Block (ACB)/Infiltration of the interspace between the popliteal artery and the capsule of the posterior knee (IPACK) versus the Periarticular Injection (PAI)/ IPACK- will be applied at the end of the surgery. dexketoprofenand paracetamol will be added to both groups and multimodal analgesia will be applied. Primary outcome is NRS pain scores with ambulation on postoperative day one (24 hours post-block administration).

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis scheduled for a primary either partial or total knee arthroplasty with a participating surgeon
* Age 18 to 80 years
* Planned use of regional anesthesia
* Ability to follow study protocol
* Patients of participating surgeons

Exclusion Criteria:

* Hepatic or renal insufficiency
* Younger than 18 years old and older than 80
* Patients undergoing general anesthesia
* Allergy or intolerance to one of the study medications
* BMI > 40
* Diabetes
* ASA of IV
* Chronic gabapentin/pregabalin use (regular use for longer than 3 months)
* Chronic opioid use (taking opioids for longer than 3 months, or daily oral morphine equivalent of >5mg/day for one month)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-12-23 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
NRS Pain Scores | 24 hours post block administration
  NRS Pain scores with ambulation 24 hours post block administration.All patients' postoperative pain numerical rating scale (NRS-numeric rating scale; 0 = absence of pain, 10 = unbearable pain) will be recorded in both groups.

SECONDARY OUTCOMES:
NRS at Rest and with movement | 24 hours on Post-Operative Day 1
  NRS at rest and with movement at different intervals. All patients' postoperative pain numerical rating scale (NRS-numeric rating scale; 0 = absence of pain, 10 = unbearable pain) will be recorded in both groups.
Patient Satisfaction with Pain Control using the likert scale | Post-Operative 24 hours
  Satisfaction with Pain control at different intervals. 1-5 (according to patient satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: Ilkay MD Baran Akkuş, MD, Principal Investigator — Diskapi Yildirim Beyazit Training Education Hospital
Locations (1):
- Diskapi Yildirim Beyazit Training Research Hospital, Ankara, Altındag, Turkey (Türkiye)